CLINICAL TRIAL: NCT04217746
Title: Effects of High Flow Nasal Cannula on Sputum Clearance in Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The pandemic interefered with the progresion of study activity.
Sponsor: Tufts Medical Center (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#13356
Record Dates: First submitted 2019-12-16; First posted 2020-01-03 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD Exacerbation; Airflow Obstruction
Keywords: high flow nasal cannula; sputum; clearability; wetability; chronic obstructive pulmonary disease; COPD exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High flow nasal cannula (HFNC) group (Experimental): The HFNC group will receive heated (approximately 37 ⁰C) and humidified (100% relative humidity) oxygenated gas delivered at high flow at 50L/min. Flow could be decreased to as low as 30L/min and temperature to 31 ⁰C as per patient's tolerance.
  Interventions: Device: High Flow Nasal Cannula
- Conventional flow nasal oxygen (CFNO) group (No Intervention): The conventional flow nasal oxygen (CFNO) group is the control group which will receive ambient temperature and non-humidified oxygen delivered at flow rates of up to 8L/min (standard care).

INTERVENTIONS:
Device: High Flow Nasal Cannula — The HFNC group will receive heated and humidified oxygenated gas delivered at high flow.
  Other Names: Fisher and Paykel AIRVO humidified high flow system
  Arms: High flow nasal cannula (HFNC) group

SUMMARY:
Acute exacerbation of COPD usually presents with more sputum production leading to worsening airflow obstruction. Often patients complain of sensation of sputum (phlegm) stuck in throat, which leads to worsening cough and respiratory distress. In an acute exacerbation setting high flow nasal cannula (HFNC), which is a modality that provides humidified and warm oxygenated air at flow of upto 60L/min, has shown to reduce blood carbon dioxide level and respiratory rate. However, studies investigating other effects of HFNC in this setting are lacking. To investigators' knowledge, this is the first study investigating effects of HFNC on sputum clearance in COPD patients.

The purpose of the study is to determine the effects of HFNC on sputum clearance in acute exacerbation of COPD. Primary objective of the study is to determine whether HFNC improves clearability and wettability of sputum produced during acute exacerbation of COPD. Secondary objectives of the study include subjective assessment of cough severity as well as need for escalation of care after HFNC use versus conventional flow nasal oxygen (CFNO) use.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of morbidity and the 4th leading cause of mortality in the world. Acute exacerbation of COPD usually presents with more sputum production leading to worsening airflow obstruction. During an exacerbation, high flow nasal cannula (HFNC) has shown to reduce blood carbon dioxide level and respiratory rate. However, studies investigating other effects of HFNC in this setting are lacking. To investigators' knowledge, this is the first study investigating effects of HFNC on sputum clearance in COPD patients.

Patients with a diagnosis of acute exacerbation of COPD who are receiving oxygen therapy via conventional nasal cannula or are on room air will be randomized into high flow nasal cannula (HFNC) or conventional flow nasal oxygen (CFNO) group for 24 hours. HFNC group will receive heated (approximately 37 ⁰C) and humidified (100% relative humidity) oxygenated gas delivered at high flow at 50L/min. CFNO group will receive ambient temperate and non-humidified oxygenated gas delivered at flow of up to 8L/min (standard care). Sputum sample will be collected at time = 0 hours (baseline), 4 +/- 1 hours, 8 +/- 2 hours and 24 +/- 2 hours. Visual analogue score (VAS) regarding cough severity and Breathlessness, Cough and Sputum Scale (BCSS) regarding cough frequency and ease will be obtained at time = 0 and 24 hours.

Primary outcomes of the study are the difference in clearability and wettability of sputum sample. Clearability is measured by the distance sputum sample travels in an artificial trachea after a simulated cough. The longer the displacement, the more the clearability. Wetability is measured by determining the contact angle the sputum sample makes on a glass surface. The smaller the contact angle, the more the wettability. Secondary outcomes include subjective assessment of cough using VAS and BCSS scales, as well as need for escalation of care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Known COPD or high probability of the disease according to treating physician based on clinical history, physical examination and chest imaging.
3. Hospital admission for acute exacerbation of COPD defined by 2018 GOLD report as acute worsening of respiratory symptoms (more than baseline cough, sputum purulence or volume, dyspnea or wheeze) that result in additional therapy.
4. Presence of one or more of following: increase in sputum production, change in sputum color or difficulty in expectorating sputum.

Exclusion Criteria:

1. Inability to obtain informed consent from the patient or legally authorized representative.
2. Inability of the subject to cooperate with protocol.
3. Presence of idiopathic bronchiectasis or cystic fibrosis.
4. Patients with poor short term prognosis not expected to survive the hospitalization.
5. Massive hemoptysis.
6. Patients presenting with coma (Glasgow coma scale <10) or circulatory shock.
7. Respiratory failure requiring non-invasive ventilation (NIV) or endotracheal intubation.
8. Severely impaired cough, impaired swallowing or chronic aspiration due to neuromuscular disorder.
9. Facial deformity or injury leading to difficulty in wearing high flow nasal cannula appropriately.
10. Enrollment in other investigative protocols with apparent overlap.
11. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Clearability of sputum sample at baseline | Sputum sample will be collected at time = 0 hours (baseline)
  Clearability is measured by the distance sputum sample travels in an artificial trachea after a simulated cough. The longer the displacement, the more the clearability.
Clearability of sputum sample at 6 hours | Sputum sample will be collected at time = 6 +/- 2 hours
  Clearability is measured by the distance sputum sample travels in an artificial trachea after a simulated cough. The longer the displacement, the more the clearability.
Clearability of sputum sample at 24 hours | Sputum sample will be collected at time = 24 +/- 2 hours
  Clearability is measured by the distance sputum sample travels in an artificial trachea after a simulated cough. The longer the displacement, the more the clearability.
Wettability of sputum sample at baseline | Sputum sample will be collected at time = 0 hours (baseline)
  Wetability is measured by determining the contact angle the sputum sample makes on a glass surface. The smaller the contact angle, the more the wettability.
Wettability of sputum sample at 6 hours | Sputum sample will be collected at time = 6 +/-2 hours
  Wetability is measured by determining the contact angle the sputum sample makes on a glass surface. The smaller the contact angle, the more the wettability.
Wettability of sputum sample at 24 hours | Sputum sample will be collected at time = 24 +/-2 hours
  Wetability is measured by determining the contact angle the sputum sample makes on a glass surface. The smaller the contact angle, the more the wettability.

SECONDARY OUTCOMES:
Change in cough severity | Visual analogue score regarding cough severity will be obtained at time = 0 hours (baseline), and time = 24 hours.
  Subjective assessment of change in cough severity using a 0mm to 100mm visual analogue scale (VAS) with 0mm being no cough to 100mm being worse cough ever.
Change in cough frequency and easiness | Breathlessness, Cough and Sputum Scale (BCSS) regarding cough frequency and ease will be obtained at time = 0 hours (baseline), and time = 24 hours.
  Subjective assessment of cough frequency and easiness using Breathlessness, Cough and Sputum Scale (BCSS) with score ranging from 0 to 12, 0 being no cough, no difficulty breathing and no trouble due to sputum and 12 being severe difficulty breathing, constant cough and constant trouble due to sputum.
Number of participants with need for escalation of care | Need for escalation will be documented at any time throughout subject's participation which is upto 24 hours.
  Need for escalation of care including non-invasive ventilation (NIV), endotracheal intubation or transfer to higher level of care.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hill, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share IPD.